CLINICAL TRIAL: NCT00602498
Title: A Single Dose, Two-Treatment, Two-Period, Two-Sequence Crossover Bioequivalency Study of 500 mg Clarithromycin Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Clarithromycin Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Director, Drug Regulatory Affairs and Medical Affairs, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 461-08
Record Dates: First submitted 2007-09-20; First posted 2008-01-28 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Infection
MeSH Terms: conditions — Infections | interventions — Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Clarithromycin

SUMMARY:
The objective of this study was the bioequivalence of a potential generic 500 mg clarithromycin tablet formulation compared with Abbott Laboratories 500 mg clarithromycin tablet, Biaxin® following a single 500 mg dose, administered with food.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening.

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C.
* Treatment with known enzyme altering drugs.
* History of allergic or adverse response to clarithromycin or any other macrolide antibiotic.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2003-03; Primary Completion 2003-03 (Actual); Study Completion 2003-03 (Actual)

PRIMARY OUTCOMES:
Bioequivalence | Baseline, Two period, Seven day washout

CONTACTS AND LOCATIONS:
Overall Officials: Irving E Weston, MD, Principal Investigator — MDS Pharma Services
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States